CLINICAL TRIAL: NCT03182205
Title: Autonomic and Hemodynamic Responses to Inspiratory Muscle Exercise in Pre Hypertensive and Hypertensive Individuals: a Randomized Clinical Trial
Brief Title: Autonomic and Hemodynamic Responses to Inspiratory Muscle Exercise in Pre Hypertensive and Hypertensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Lilian Pinto da Silva, Autonomic and Hemodynamic Responses to Inspiratory Muscle Exercise in Pre Hypertensive and Hypertensive Individuals, Federal University of Juiz de Fora
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAE64969617000005133
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Prehypertension; Hypertension
Keywords: Breathing Exercises; Autonomic Nervous System; Hemodynamics
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle exercise (IME) (Experimental): Participants will be submitted to a linear pressure resistance (PowerBreathe) with an inspiratory load of 40% of maximal inspiratory pressure.
  Interventions: Other: IME
- Sham IME (Sham Comparator): Participants will be submitted to inspiratory muscle exercise with the same equipment as the intervention group, but without a load generating resistance.
  Interventions: Other: Sham IME

INTERVENTIONS:
Other: IME — The IME session protocol will consist of 8 sets of 2 minutes with 1 minute rest between sets. Inspiratory load will be set at 40% of maximum static inspiratory pressure. In addition, the volunteer will be instructed to perform diaphragmatic breathing, maintaining a respiratory rate in the range of 12 to 15 ipm (feedback from the evaluator) and the entire exercise protocol will be performed with the patient sitting with their feet flat on the floor and using a clip nasal.
  Other Names: Inspiratory muscle exercise
  Arms: Inspiratory muscle exercise (IME)
Other: Sham IME — The Sham IME session protocol will consist of 8 sets of 2 minutes with 1 minute rest between sets, but without a load generating resistance. In addition, the volunteer will be instructed to perform diaphragmatic breathing, maintaining a respiratory rate in the range of 12 to 15 ipm (feedback from the evaluator) and the entire exercise protocol will be performed with the patient sitting with their feet flat on the floor and using a nasal clip.
  Other Names: Sham inspiratory muscle exercise
  Arms: Sham IME

SUMMARY:
This study aims to evaluate the autonomic and hemodynamic responses triggered by inspiratory muscle exercise in prehypertensive and hypertensive individuals. The reason that leads us to this study refers to clinical relevance for individuals with high blood pressure levels, since this type of exercise can act as a important nonpharmacological agent for arterial pressure control. In addition, this study aims to elucidate the mechanisms involved in cardiovascular responses to inspiratory muscle exercise and, consequently, provide safety in the prescription of these for this population.

DETAILED DESCRIPTION:
This is a randomized clinical trial, consisting of a convenience sample of patients from the Cardiology Department of the University Hospital (UH) of the Federal University of Juiz de Fora (FUJF). The patients will be invited to participate in the study and will receive information regarding the objectives and procedures of the study. In case of agreement with their inclusion in the study, they will sign a free and informed consent form.

The entire experiment will be carried out in the Physical Evaluation Laboratory of the UH-FUJF, by the researchers previously trained in the application of the protocol. The stages of the experimental protocol will be divided into three days as described below.

1. 1st day of the experimental protocol (initial evaluation): medical historical, anthropometric evaluation, electrocardiographic monitoring at rest, evaluation of respiratory muscle strength and familiarization with the muscle training device. All volunteers will be instructed to refrain from taking caffeinated and alcoholic beverages for 24 h before the evaluation and to have a good night's sleep.
2. 2nd and 3rd days of the experimental protocol: all volunteers will be randomly assigned to two exercise sessions (ES): Sham IME (no load) and moderate intensity IME (40% of MIP). Initially, the volunteers will perform a 10-minute supine rest for heartbeat collection and subsequent calculation of heart rate variability (HRV), blood pressure and forearm blood flow measurements and evaluation of the baroreflex system. In sequence the ES will be conducted with continuous monitoring of blood pressure, heart rate and subjective perception of effort through the Borg Scale. Immediately and until one hour after the ES, it will be measured forearm blood flow, blood pressure, heart rate and evaluated the baroreflex system and HRV in order to investigate the acute effect of ES. The volunteers will be monitored using an equipment capable of evaluating the outpatient measurement of blood pressure and electrocardiogram for 24 hours in order to investigate the chronic effect of ES.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of prehypertension (systolic blood pressure > 121-139 mmHg / diastolic blood pressure > 81-89 mmHg) and stage 1 hypertension (systolic blood pressure > 140-159 mmHg / diastolic blood pressure > 90-99 mmHg) with low to moderate cardiovascular risk
* Do not use drugs to control blood pressure levels
* Sedentary for at least 6 months

Exclusion Criteria:

* Cardiovascular or respiratory diseases
* Arrhythmias detected during electrocardiographic monitoring
* Inability to perform the proposed protocol

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood pressure levels in 24 hours | Baseline, 60 minutes and 24 hours post each intervention
  Noninvasive hemodynamic monitoring and ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Autonomic nervous system | Baseline, 60 minutes and 24 hours post each intervention
  Heart rate variability
Peripheral blood flow | Baseline and 60 minutes post each intervention
  Plethysmography of venous occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Lilian P Silva, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Hospital Universitário da UFJF, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archiza B, Simoes RP, Mendes RG, Fregonezi GA, Catai AM, Borghi-Silva A. Acute effects of different inspiratory resistive loading on heart rate variability in healthy elderly patients. Braz J Phys Ther. 2013 Jul-Aug;17(4):401-8. doi: 10.1590/S1413-35552012005000100. Epub 2013 Aug 23. PMID 23970114
- [Background] Ferreira JB, Plentz RD, Stein C, Casali KR, Arena R, Lago PD. Inspiratory muscle training reduces blood pressure and sympathetic activity in hypertensive patients: a randomized controlled trial. Int J Cardiol. 2013 Jun 5;166(1):61-7. doi: 10.1016/j.ijcard.2011.09.069. Epub 2011 Oct 9. PMID 21985749
- [Background] Hering D, Kucharska W, Kara T, Somers VK, Parati G, Narkiewicz K. Effects of acute and long-term slow breathing exercise on muscle sympathetic nerve activity in untreated male patients with hypertension. J Hypertens. 2013 Apr;31(4):739-46. doi: 10.1097/HJH.0b013e32835eb2cf. PMID 23385649
- [Background] McConnell AK, Griffiths LA. Acute cardiorespiratory responses to inspiratory pressure threshold loading. Med Sci Sports Exerc. 2010 Sep;42(9):1696-703. doi: 10.1249/MSS.0b013e3181d435cf. PMID 20142783
- [Background] Ramos PS, Da Costa Da Silva B, Gomes Da Silva LO, Araujo CG. Acute hemodynamic and electrocardiographic responses to a session of inspiratory muscle training in cardiopulmonary rehabilitation. Eur J Phys Rehabil Med. 2015 Dec;51(6):773-9. Epub 2015 Feb 5. PMID 25653080
- [Background] Rodrigues F, Araujo AA, Mostarda CT, Ferreira J, de Barros Silva MC, Nascimento AM, Lira FS, De Angelis K, Irigoyen MC, Rodrigues B. Autonomic changes in young smokers: acute effects of inspiratory exercise. Clin Auton Res. 2013 Aug;23(4):201-7. doi: 10.1007/s10286-013-0202-1. Epub 2013 Jun 28. PMID 23812534
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284